CLINICAL TRIAL: NCT01100099
Title: HLA-DQ2-gliadin Tetramer for Diagnosis of Celiac Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: South-Eastern Norway Regional Health Authority (Other); University of Oslo (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2007068; 2007068 2009021 (Other: Health Administration of Eastern Norway)
Record Dates: First submitted 2010-04-06; First posted 2010-04-08 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2012-09

CONDITIONS: Celiac Disease; Gluten
Keywords: Celiac disease.; Food intolerance.; Gluten intolerance without celiac disease.
MeSH Terms: conditions — Celiac Disease; Food Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gluten challenge. (Experimental): Diagnosis of celiac disease. Before and after a gluten challenge small bowel biopsies will be taken, and blood samples will be drawn for tetramer staining of gluten specific T cells.
  Interventions: Dietary Supplement: Gluten challenge.

INTERVENTIONS:
Dietary Supplement: Gluten challenge. — The study population consists of 50 HLA-DQ2+ patients on a gluten free diet, both celiacs and uncertain celiacs. The patients will undergo a oral gluten challenge with four slices of bread daily for three days. Before challenge blood samples will be drawn for tetramer staining of gluten-specific T-cells. The analysis is done at the Institute of Immunology at Rikshospitalet, using FACS analysis. Small intestinal biopsies will be examined for morhological changes and inflammatory gene expression. These procedures with blood samples and biopsies will be repeated after gluten challenge. Registration for clinical symptoms and personality traits will be done by standardised and validated forms. A dietist will perform an interview of the patients.

SUMMARY:
The investigators will evaluate the use of an HLA-DQ2-gliadin tetramer for staining of gluten specific T cells in the diagnostics of uncertain celiac disease. Some patients have started on a gluten free diet without a diagnosis of celiac disease. Subsequent later investigation in special care is difficult as the patients often are reluctant to prolonged gluten challenge. The investigators use the HLA-DQ2-gliadin tetramers for detection of gluten specific T cells after a short gluten challenge. By this method the investigators search to discriminate between true celiac disease and clinical gluten intolerance without celiac disease, in a population of HLA-DQ2+ persons already on a gluten free diet without a formal diagnosis of celiac disease.

ELIGIBILITY:
Inclusion Criteria:

* HLA-DQ2+ celiacs and HLA-DQ2+ persons who have been on a gluten free diet for at least 4 weeks.

Exclusion Criteria:Pregnancy

* Other severe disease
* Refusal to participate
* HLA-DQ2 negativity

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-09; Primary Completion 2009-12 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
HLA-DQ2-tetramer response after gluten challenge | 6 days.
  FACS analysis of peripheral blood after gluten challenge.

SECONDARY OUTCOMES:
Mucosal responses to 3 day gluten challenge. | 4 days.
  Biopsy the fourth day of gluten challenge.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine, Endoscopy Unit, Rikshospitalet, Oslo, Norway

REFERENCES:
- [Background] Raki M, Fallang LE, Brottveit M, Bergseng E, Quarsten H, Lundin KE, Sollid LM. Tetramer visualization of gut-homing gluten-specific T cells in the peripheral blood of celiac disease patients. Proc Natl Acad Sci U S A. 2007 Feb 20;104(8):2831-6. doi: 10.1073/pnas.0608610104. Epub 2007 Feb 16. PMID 17307878